CLINICAL TRIAL: NCT05983874
Title: An Open-Label Study to Evaluate the Safety and Immunogenicity of 2 Doses of 100µg BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, Given to a Population of Adults in Good General Health Who Have Received 3 Doses of 300µg BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted
Brief Title: A Study to Evaluate the Safety and Immunogenicity of 2 Doses of 100µg BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, Given to a Population of Adults Who Have Received 3 Doses of 300µg BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: 3M (Industry); Access to Advanced Health Institute (AAHI) (Other); Polymun Scientific GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IAVI C110
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — aluminum sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1: BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) Dosage (Experimental): BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum)
  Interventions: Biological: BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) Dosage

INTERVENTIONS:
Biological: BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) Dosage — 100µg Month 0 and Month 3

SUMMARY:
An Open-Label Study to Evaluate the Safety and Immunogenicity of 2 Doses of 100µg BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, given to a Population of Adults in Good General Health Who have Received 3 doses of 300µg BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted

DETAILED DESCRIPTION:
The study population is comprised of adults in good general health who meet all protocol inclusion criteria and do not meet any protocol exclusion criteria and who understand the study and provide written informed consent.

Up to 8 participants who received 3 doses of 300µg of BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted, from the AMC clinical site in IAVI C101 (NCT04224701) will be enrolled in the study.

BG505 SOSIP.664 gp140 is a stable, soluble, cleaved HIV envelope trimer formulated in 0.55mL at 2mg/mL in 20 mM Tris, 100mM Sodium Chloride (NaCl), pH 7.5 and will be administered intramuscular (IM).

BG505 SOSIP.664 gp140 will be diluted in 20 mM Tris, 100 mM NaCl, pH 7.5 (Tris NaCl Diluent).

The 3M-052-AF is provided by AAHI. 3M-052-AF is provided in 2mL vials, with a fill volume of 0.4mL at a concentration of 50µg/mL. 3M 052 AF is a clear-to-slightly hazy, colorless liquid.

Aluminum hydroxide suspension 2% is a pyrogen free, sterilized aluminum hydroxide wet gel suspension, placed into 2 mL Type 1 vials, containing an aluminum concentration of 10 mg/mL. It appears as an opaque white gelatinous precipitate in aqueous suspension.

All administrations of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted will be given IM in a 0.5mL volume. The study product is described in detail in the Investigators Brochure.

All products slated for use in the Netherlands will have EU-compliant labels.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults as assessed by a medical history, physical exam, and laboratory tests
2. Received 3 doses of 300µg of BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted
3. Willing to comply with the requirements of the protocol and be available for follow-up for the planned duration of the study
4. In the opinion of the Principal Investigator (PI), or designee, and based on Assessment of Understanding (AOU) results, has understood the information provided and potential impact and/or risks linked to vaccine administration and participation in the trial; written informed consent will be obtained from the participant before any study-related procedures are performed
5. Willing to undergo HIV testing, risk reduction counseling and receive HIV-test results
6. All participants born female who are engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception starting 2 weeks before the first vaccine administration and for 4 months following the last vaccine administration. Effective contraception includes:

   * Condoms (male or female) with or without spermicide
   * Diaphragm or cervical cap with spermicide
   * Intrauterine device
   * Hormonal contraception, including contraceptive implant or injectable
   * Oral contraception
   * Successful vasectomy in the male partner

Considered successful if a woman reports that a male partner has:

1. documentation of azoospermia by microscopy (1 year ago) or
2. a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post vasectomy • Not of reproductive potential Such as having undergone hysterectomy, bilateral oophorectomy, or tubal ligation, postmenopausal (≥45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level > 40 IU/L), surgically sterile Note: More restrictive measures may be required by the study sites. 7. All participants born female who are not heterosexually active at screening must agree to utilize an effective method of contraception if they become heterosexually active as outlined above 8. All participants born female must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Assessments (SOA) (Appendix A) 9. Willing to forgo donations of blood, or any other tissues during the study and, for those who test HIV-positive due to vaccine-induced antibodies, until the anti-HIV-antibody titers become undetectable 10. For sites in the European Union (EU), participant consents to the collection and use of personal data in compliance with the General Data Protection Regulation

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection
2. Any clinically relevant abnormality on history or examination, including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical or inhaled steroids is permitted), immunosuppressive, anticancer, anti-tuberculosis or other medications considered significant by the Investigator within the previous 6 months.

   Note: The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on Investigator clinical judgment) at least 2 weeks prior to enrollment in this study.
3. Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the Investigator makes the participant unsuitable for participation in the study
4. Reported behavior that put the participant at risk for HIV infection within 6 months prior to vaccine administration, as defined by:

   * Unprotected sexual intercourse with a known HIV-infected person, a partner known to be at high risk for HIV infection or a casual partner (ie, no continuing established relationship)
   * Engaged in sex work
   * Frequent excessive daily alcohol use or frequent binge drinking, or any other use of illicit drugs
   * History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, HSV-2, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B or hepatitis C
   * Three or more sexual partners
5. If female, pregnant, lactating, or planning a pregnancy during the period of enrollment until 4 months after the last vaccine administration
6. Bleeding disorder that was diagnosed by a physician (eg, clotting factor deficiency, coagulopathy or platelet disorder that requires special precautions) Note: A participant who states that he/she has easy bruising or bleeding, but does not have a formal diagnosis and has IM injections and blood draws without any adverse experience is eligible
7. Infectious disease diagnosis: chronic hepatitis B infection (HbsAg-positive), current hepatitis C infection (HCV Ab positive and HCV ribonucleic acid (RNA) positive or interferon-alfa treatment for hepatitis C infection in the past year or interferon-alfa-free treatment for hepatitis C infection completed in the past 6 months), or active syphilis (screening and confirmatory tests)
8. History of splenectomy
9. Any of the following abnormal laboratory parameters listed below:

   Hematology
   * Hemoglobin - <10.5 g/dl or <6.5 mmol/L in females; <11.0 g/dl or <6.8 mmol/L in males
   * Absolute Neutrophil Count (ANC) - ≤1,000/mm3 or < 1.0 x 109 cells/L
   * Absolute Lymphocyte Count (ALC) - ≤650/mm3 or < 0.65 x 109 cells/L
   * Platelets - <125,000 cells/mm3 or <125 x 109 cells/L Chemistry
   * Creatinine - >1.1 x upper limit of normal (ULN)
   * AST - >1.25 x ULN
   * ALT - >1.25 x ULN Urinalysis

   Clinically significant abnormal dipstick confirmed by microscopy:
   * Protein = 1+ or more
   * Blood = 2+ or more (not due to menses)
10. Receipt of live attenuated vaccine within the previous 30 days or planned receipt within 30 days after vaccine administration; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after vaccine administration. (Exception is live attenuated influenza vaccine within 14 days.)
11. Receipt of blood transfusion or blood-derived products within the previous 3 months
12. Participation in another clinical trial of a vaccine currently, within the previous 3 months or expected participation during this study (with the exception of Protocol IAVI C101); concurrent participation in an observational trial not requiring blood or tissue sample collection is not an exclusion
13. Prior receipt of any investigational HIV vaccine candidate or HIV monoclonal antibody other than BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted
14. History of significant local or systemic reactogenicity to vaccines (eg, anaphylaxis, respiratory difficulties, angioedema, injection site necrosis or ulceration)
15. Psychiatric condition that compromises safety of the participant and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
16. Seizure disorder: A participant who has had a seizure in the last 3 years is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years)
17. History of malignancy in the past 5 years (prior to screening) or ongoing malignancy (a history of completely excised malignancy, which is considered cured, is not an exclusion)
18. Active, serious infections requiring antibiotic, antiviral, or antifungal therapy within 30 days prior to enrollment
19. Body mass index (BMI) ≥35
20. Body weight <110 pounds (50 kg)
21. Prior daily use of NSAID/aspirin that cannot be held for 5 days prior to the leukapheresis procedure (if required by the study site)
22. If, in the opinion of the PI, it is not in the best interest of the participant to participate in the trial

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Grade 2 or greater reactogenicity (ie, solicited AEs) from Day 0 through Day 7 after each vaccine administration | 7 days
Proportion of participants with vaccine-related unsolicited AEs, including safety laboratory (biochemical, hematological) parameters, from the day of each vaccine administration up to 28 days post each vaccine administration | 28 days
Proportion of participants with Grade 2 or greater unsolicited AEs, including safety laboratory (biochemical, hematological) parameters, from the day of each vaccine administration up to 28 days post each vaccine administration | 28 days
Proportion of participants with vaccine-related SAEs throughout the study period | 7 months
Proportion of participants in each group with potential immune-mediated diseases (pIMDs) from the day of first vaccine administration throughout the study period | 7 months

SECONDARY OUTCOMES:
Frequency and magnitude of binding antibody responses to 2 doses of 100µg of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, given to adults in good general health who have received 3 doses of 300ug of BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Godelieve de Bree, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- The Amsterdam University Medical Centers, Amsterdam, Netherlands